CLINICAL TRIAL: NCT04539743
Title: Modified Step by Step Mitrofanoff Continent Cystostomy : Functional Results of a Teachable Procedure
Acronym: MCCR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.193; 2020-A0156534 (Other: ID RCB)
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Mitrofanoff Continent Cystostomy; Cystostomy; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The creation of an abdominal continental cystostomy orifice is an irreplaceable surgical technique that allows for the simple self-sounding of the bladder in patients with severe disabilities or malformations, and to obtain urinary continence.

This operation, the principle of which was described by Paul Mitrofanoff in 1980, has benefited from countless descriptions, difficult realization and questionable design, so it is insufficiently proposed.

Faced with this learning difficulty at the beginning of the year, we decided to define a "step-by-step" technique, in seven well-differentiated steps. This approach has simplified the teaching and dissemination of this technique.

To validate its quality, it is necessary to evaluate the expected results of a continental cystostomy, by answering two simple questions:

-is the cystostomy opening really continent? Is the cystostomy tube easy to catheterize?

DETAILED DESCRIPTION:
This research consists in highlighting that the Mitrofanoff surgery technique used by the CHUGA surgeons during a cystostomy is easier to perform while having the necessary same results as the other methods.

To do this, we must validate the quality of this method and therefore we will evaluate the results expected from a continuous cystostomy via a questionnaire. After a first telephone contact by Dr BOILLOT for a presentation of the study, patient will therefore be contacted by telephone by the Clinical Research Associate of the service.

During this interview patient will be asked to answer a questionnaire consisting of five questions.

ELIGIBILITY:
Inclusion Criteria:

* adult who has undergone a Mitrofanoff cystostomy by Dr. BOILLOT

Exclusion Criteria:

* Persons referred to in Articles L1121-5 to L1121-8 of the CSP (corresponds to all protected persons: pregnant women, parturient women, nursing mothers, persons deprived of their liberty by judicial or administrative decision, persons subject to a legal protection measure)
* Patients operated on by other surgeons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult who has undergone a Mitrofanoff cystostomy by Dr. BOILLOT
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate, in a series of identically operated patients, the expected results of a continuous cystostomy: -is the cystostomy hole really continental? -is the cystostomy tube easy to catheterize | 1 month
  Average of the Scores obtained on the questionnaires carried out

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Grenoble Alpes, Grenoble, France